CLINICAL TRIAL: NCT02751177
Title: Multicenter Prospective Study Comparing KRAS, NRAS and BRAF Mutation Testing Using OncoBEAM Technique in Plasma vs Conventional Techniques in Formalin Fixed Paraffin Embedded Tissues
Brief Title: Detection of KRAS, NRAS et BRAF Mutations in Plasma Circulating DNA From Patients With Metastatic Colorectal Cancer
Acronym: ColoBEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A01272-47
Record Dates: First submitted 2016-03-03; First posted 2016-04-26 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer Metastatic
Keywords: KRAS gene mutation; NRAS gene mutation; BRAF gene mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OncoBEAM (Experimental): KRAS, NRAS and BRAF mutations will be analyzed in circulating plasma DNA using ONCOBEAM technique.
  Interventions: Genetic: KRAS, NRAS et BRAF mutation analysis from circulating plasma DNA

INTERVENTIONS:
Genetic: KRAS, NRAS et BRAF mutation analysis from circulating plasma DNA — Mutation in plasma DNA vs tumor tissue
  Other Names: metastatic colorectal cancer; OncoBEAM

SUMMARY:
RAS genotyping is mandatory for the prescription of anti-EGFR (epidermal growth factor receptor) therapies in patients with metastatic colorectal cancer. The standard genotyping is assessed on formalin-fixed paraffin embedded tumour tissue. This study compares RAS and BRAF genotyping results achieved in analyzing circulating plasma DNA using OncoBEAM™ technique with those achieved using the standard genotyping techniques and formalin-fixed paraffin embedded samples.

DETAILED DESCRIPTION:
The study will be proposed to all patients with a metastatic colorectal cancer.

Study information will be given to the patient during a routine medical examination. The patient will be included after checking inclusion criteria and signature of the informed consent form

Blood sampling (30 ml) will be performed before the initiation of the first line metastatic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with newly diagnosed, anti EGFR treatment naïve metastatic colorectal cancer
* Standard of Care RAS/RAF tests performed on FFPE tumor sample as part of routine
* Patient information and written informed consent form signed
* Patient must be affiliated to a social security system
* Age : 18 years and older

Exclusion Criteria:

* Patient bearing non-metastatic colorectal cancer
* Patient with local relapse only
* Patient with exclusive nodal metastases
* Patient whose health contraindicates a 30 ml blood sample
* Blood transfusion within 1 week prior blood collection
* Patient having received any chemotherapy or / and radiotherapy within 15 days prior to blood collection
* History of another primary cancer within the last 5 years, with the exception of non-melanomatous skin cancer and carcinoma in situ of the cervix
* Persons deprived of liberty or under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
KRAS, NRAS et BRAF mutational status | up to 6 months
  Compare the results of KRAS (exons 2, 3 et 4), NRAS (exons 2, 3 et 4) and BRAF (V600) genes genotyping using OncoBeam technique in blood samples with results achieved routinely by the molecular genetics platforms of the recruiting centers.

CONTACTS AND LOCATIONS:
Overall Officials: MERLIN JEAN LOUIS, Study Chair — Institut de Cancérologie de Lorraine; HARLE ALEXANDRE, Study Chair — Institut de Cancérologie de Lorraine; GAVOILLE CELINE, oncologist, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (11):
- France (11):
  - CH Auxerre, Auxerre
  - CH Besançon-Hopital Jean Minjoz, Besançon
  - CH Chalon Sur Saône-William Morey, Chalon-sur-Saône
  - Centre Georges François Leclerc Dijon, Dijon
  - Hopital Belle-Isle-Metz, Metz
  - Polyclinique de Gentilly, Nancy
  - CHU Reims-Hôpital Robert Debré, Reims
  - Polyclinique Courlancy Reims, Reims
  - Centre Paul Stauss, Strasbourg
  - CHRU Nancy, Vandœuvre-lès-Nancy
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Harle A, Gavoille C, Bouche O, Abdelghani MB, Plaza J, Spaeth D, Boudrant A, Ghiringhelli F, Villing AL, Borg C, Rouyer M, Husson M, Gilson P, Salleron J, Lambert A, Merlin JL. Sensitive cell-free DNA assay for accurate detection of RAS and BRAF mutations in liquid biopsies of patients with metastatic colorectal cancer: Final results of the multicentric ColoBEAM study. Oncol Lett. 2025 Oct 30;31(1):13. doi: 10.3892/ol.2025.15366. eCollection 2026 Jan. PMID 41235357